CLINICAL TRIAL: NCT02485561
Title: Comparing Screener vs. Survivor Role Models to Improve Colon Cancer Screening
Brief Title: Evaluating Strategies to Present Colon Cancer Screening Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amy McQueen, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HRPO201501019; R21CA187608 (NIH)
Record Dates: First submitted 2015-06-18; First posted 2015-06-30 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Colonic Neoplasms; Colorectal Neoplasms; Colonic Diseases; Gastrointestinal Neoplasms
Keywords: Colon cancer screening; Colorectal cancer screening; Colonoscopy; Sigmoidoscopy; Stool blood test; Narrative
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Colonic Diseases; Gastrointestinal Neoplasms; Narration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Information only (Active Comparator): INTERVENTION: Information about colon cancer and screening tests from sources such as the Centers for Disease Control and Prevention Screen for Life campaign.
  Interventions: Behavioral: Education information
- Screener Narrative (Experimental): INTERVENTION: Information + Personal Narrative from someone who was screened for colon cancer
  Interventions: Behavioral: Health communication intervention; Behavioral: Education information
- Survivor Narrative (Experimental): INTERVENTION: Information + Personal Narrative from someone who was screened for, and diagnosed with, colon cancer
  Interventions: Behavioral: Health communication intervention; Behavioral: Education information

INTERVENTIONS:
Behavioral: Health communication intervention — This study will compare the effects of adding narratives that describe personal experiences with colon cancer screening to educational information alone to explore potential differences in reactions to different role models on individuals' screening intentions and behaviors.
  Arms: Screener Narrative; Survivor Narrative
Behavioral: Education information — Educational materials such as those from the Centers for Disease Control and Prevention are used to present educational information to participants about colon cancer and screening tests.

SUMMARY:
This is a study examining the effects of different educational-motivational materials about colorectal cancer screening on perceptions and intentions to get screened. Eligible participants will be randomized to one of three experimental conditions. All participants will be provided information about colon cancer and screening options based on the Centers for Disease Control and Prevention Screen for Life materials. Some participants also will be asked to read a personal narrative about colon cancer screening. This study will determine whether participant's perceptions about and colorectal cancer screening intentions and behaviors differ by which information they read. Participants will complete surveys before, immediately after, and one month after randomization. To assess behavior change, as suggested by grant reviewers and the project officer, we added 6 and 12 month follow up surveys. Participants can complete all study requirements through the study website: http://HealthStudy.wustl.edu

DETAILED DESCRIPTION:
The use of patient narratives in interventions and their availability on the Internet is becoming ubiquitous and has far outpaced empirical research to assess how and for whom narratives are effective. To improve future behavioral interventions that incorporate narratives, researchers need to identify the best role models to promote colon cancer screening and examine their potentially different mechanisms of influence.

For the proposed web-based, 3-arm English-language pilot intervention with a brief, 1 month follow-up, the study investigators will randomize 400 average-risk adults age 50-75 who are non-adherent to colon cancer screening guidelines and have no cancer history to one of three groups to read: 1) basic information about colon cancer risk and test options, 2) the same colon cancer and screening information plus a narrative from a colon cancer survivor, or 3) the same colon cancer and screening information plus a narrative from someone who got screened for colon cancer. To better assess behavior change, a 6 and 12 month follow up survey was added.

All participants will read general information about colon cancer and screening guidelines, test options, and benefits based on Centers for Disease Control and Prevention educational materials. Narrative participants will then view a role model that is tailored to each participant by gender, race/ ethnicity, and age group. Along with a photo will be a brief message to identify role models as colon cancer survivors or screeners. Narrative conditions will include a single role model and story of first-person experiences of colonoscopy. Participants will complete survey measures before and after the information and stories are presented and at one, 6, and 12 month follow-up. Participation in the first part of the study will take about 30 minutes and about 15 minutes for the follow up survey. Participants can complete all study requirements through our website: http://HealthStudy.wustl.edu

This study will examine potential mediators or mechanisms that explain the effects of these narratives on screening-related outcomes based on a proposed conceptual model. The study investigators will enroll a diverse sample of participants to explore any differences in narrative effects by audience characteristics (potential moderators).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults of any race or ethnicity living in the United States
* Age 50-75 years old
* Access to the Internet to complete all study requirements at http://HealthStudy.wustl.edu

Exclusion Criteria:

* Unable to read English
* Prior diagnosis of cancer (except non-melanoma skin cancer)
* Prior diagnosis of Crohn's disease, inflammatory bowel disease or colitis
* Currently adherent to colon cancer screening guidelines defined as a home-based stool blood test in the past 12 months, a sigmoidoscopy in the past 5 years, or a colonoscopy in the past 10 years.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy McQueen, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University website HeathStudy.wustl.edu, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
A data sharing agreement with an interested researcher that complies with federal, university, and institution review board standards for protecting data.

REFERENCES:
- [Background] Weinstein ND, Kwitel A, McCaul KD, Magnan RE, Gerrard M, Gibbons FX. Risk perceptions: assessment and relationship to influenza vaccination. Health Psychol. 2007 Mar;26(2):146-51. doi: 10.1037/0278-6133.26.2.146. PMID 17385965
- [Background] Sestir M, Green MC. You are who you watch: Identification and transportation effects on temporary self-concept. Social Influence 5(4): 272-88, 2010.
- [Background] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231
- [Background] Green MC, Brock TC. The role of transportation in the persuasiveness of public narratives. J Pers Soc Psychol. 2000 Nov;79(5):701-21. doi: 10.1037//0022-3514.79.5.701. PMID 11079236
- [Background] McQueen A, Kreuter MW, Kalesan B, Alcaraz KI. Understanding narrative effects: the impact of breast cancer survivor stories on message processing, attitudes, and beliefs among African American women. Health Psychol. 2011 Nov;30(6):674-82. doi: 10.1037/a0025395. Epub 2011 Sep 5. PMID 21895370
- [Background] McQueen A, Kreuter MW. Women's cognitive and affective reactions to breast cancer survivor stories: a structural equation analysis. Patient Educ Couns. 2010 Dec;81 Suppl:S15-21. doi: 10.1016/j.pec.2010.08.015. Epub 2010 Sep 17. PMID 20850258
- [Background] McQueen A, Vernon SW, Swank PR. Construct definition and scale development for defensive information processing: an application to colorectal cancer screening. Health Psychol. 2013 Feb;32(2):190-202. doi: 10.1037/a0027311. Epub 2012 Feb 20. PMID 22353026
- [Background] McQueen A, Swank PR, Vernon SW. Examining patterns of association with defensive information processing about colorectal cancer screening. J Health Psychol. 2014 Nov;19(11):1443-58. doi: 10.1177/1359105313493649. Epub 2013 Jul 17. PMID 23864072
- [Background] McQueen A, Tiro JA, Vernon SW. Construct validity and invariance of four factors associated with colorectal cancer screening across gender, race, and prior screening. Cancer Epidemiol Biomarkers Prev. 2008 Sep;17(9):2231-7. doi: 10.1158/1055-9965.EPI-08-0176. PMID 18768488
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Vernon SW, Meissner H, Klabunde C, Rimer BK, Ahnen DJ, Bastani R, Mandelson MT, Nadel MR, Sheinfeld-Gorin S, Zapka J. Measures for ascertaining use of colorectal cancer screening in behavioral, health services, and epidemiologic research. Cancer Epidemiol Biomarkers Prev. 2004 Jun;13(6):898-905. No abstract available. PMID 15184243
- [Derived] McQueen A, Caburnay C, Kreuter M, Sefko J. Improving Adherence to Colorectal Cancer Screening: A Randomized Intervention to Compare Screener vs. Survivor Narratives. J Health Commun. 2019;24(2):141-155. doi: 10.1080/10810730.2019.1587109. Epub 2019 Mar 29. PMID 30924402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We sent electronic invitations to prospective participants from two opt-in registries: 1) Washington University's Volunteer for Health Research Participant Registry and 2) ResearchMatch.org hosted by Vanderbilt University.
Pre-assignment Details: Nearly all participants completed all study components online. They provided informed consent and proceeded to the baseline survey (n=486). Only those that completed the baseline survey were randomized (n=477) to one of three intervention conditions, so that number is smaller than the total who started the study.
Groups:
- Information Only: INTERVENTION: Information about colon cancer and screening tests.
  Education information: Typical materials are used to present educational information to participants about colon cancer and screening tests.
- Screener Narrative: INTERVENTION: Information + Personal Narrative from someone who was screened for colon cancer
  Health communication intervention: This study will compare the effects of adding personal experiences with colon cancer screening to educational information to explore potential differences in reactions to different role models on individuals' screening intentions and behaviors.
  Education information: Typical materials are used to present educational information to participants about colon cancer and screening tests.
- Survivor Narrative: INTERVENTION: Information + Personal Narrative from someone who was screened for, and diagnosed with, colon cancer
  Health communication intervention: This study will compare the effects of adding personal experiences with colon cancer screening to educational information to explore potential differences in reactions to different role models on individuals' screening intentions and behaviors.
  Education information: Typical materials are used to present educational information to participants about colon cancer and screening tests.
Period: Overall Study
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Started | 161 | 157 | 159
Completed 1 mo Survey | 145 | 138 | 144
Completed (Completed 12 month follow up survey (final time point)) | 133 | 118 | 136
Not Completed | 28 | 39 | 23

BASELINE CHARACTERISTICS:
Population: Participants who completed the baseline survey and were randomized to receive the assigned study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Information Only | Screener Narrative | Survivor Narrative | Total
Number analyzed (Participants) | 161 | 157 | 159 | 477
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (5.8) | 57.8 (6.6) | 57.4 (6.2) | 57.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 108 | 117 | 334
  Male | 52 | 49 | 42 | 143
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 123 | 126 | 128 | 377
  African American/Black | 28 | 24 | 25 | 77
  Other race | 10 | 7 | 6 | 23
Any prior colorectal cancer screening [Count of Participants; unit: Participants] — Receipt of any colorectal screening test (i.e., home stool blood test, sigmoidoscopy, colonoscopy)
  Participants | 45 | 57 | 51 | 153

OUTCOME MEASURES:

1. Primary Outcome: Intentions to Get Screened for Colon Cancer
Description: Intention was measured on all surveys with the mean of 3 items assessed using slider bars (coded 1=not at all - 100=extremely) asking about the likelihood of being screened in the next 6 months, the importance of screening, and commitment to screening. Higher scores indicate greater intentions to get screened for colorectal cancer.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline, intervention, and immediately post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a 0-100 scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a 0-100 scale | 68.64 (26.42) | 65.51 (27.29) | 64.30 (29.99)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .362, ANOVA; F-value = 1.019

2. Secondary Outcome: Identification With the Character
Description: Participants assigned to narrative conditions were asked if they liked and felt similar to the character in the story they read with 3 items each with response options 1=Strongly Disagree - 5=Strongly Agree. Measures were based on previous work by the study investigators. Mean scores for liking and similarity were created; higher scores reflect higher perceived similarity and liking for the character. Means will be compared between the two groups assigned to read a narrative.
Time Frame: Immediately post-intervention
Population: Participants who completed baseline, intervention, and immediately post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a 5-point response scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a 5-point response scale
  Perceived similarity | NA (NA) — Info only participants did not get narratives thus did not have someone to compare themselves to | 3.69 (0.81) | 3.47 (0.91)
  Liking of character | NA (NA) — Info only participants did not get narratives thus did not have someone to indicate their liking of | 3.73 (0.63) | 3.75 (0.69)
Statistical Analysis 1: Comparison: Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .024, t-test, 2 sided; Mean Difference (Final Values) = .22, Standard Error of Mean .098
Statistical Analysis 2: Comparison: Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .75, t-test, 2 sided; Mean Difference (Final Values) = -.024, Standard Error of Mean .074

3. Secondary Outcome: Three Measures of Engagement
Description: Confirmatory factor analyses did not support an aggregate measure adapted from an existing transportation scale, so a single item "What I just read affected me emotionally" was used to measure emotional engagement for all participants. For participants assigned to either narrative condition, two items reflected cognitive (imagery) engagement "While I was reading the story, I could easily picture the events in it taking place" and "I had a vivid mental image of the person in the story". Mean scores were created for cognitive engagement. Two items reflected self-referencing engagement: "I could picture myself in the scene of the events described in the story" and "The events in the story are relevant to my life" were assessed and mean scores created for self-referencing engagement. Responses for all items were 1=Not at all - 7=Very much. Higher mean scores reflected higher engagement.
Time Frame: Immediately post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a scale
  Emotional engagement | 2.95 (1.86) | 3.05 (1.80) | 3.65 (1.94)
  Cognitive engagement | NA (NA) — Info only participants were not exposed to a narrative so could not report on imagery from reading a story | 5.45 (1.35) | 5.47 (1.31)
  Self-referencing engagement | NA (NA) — Info only participants were not exposed to a narrative so could not report on how the story relates to themselves | 5.23 (1.47) | 4.51 (1.73)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .002, ANOVA; F-value = 6.482
Statistical Analysis 2: Comparison: Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .91, t-test, 2 sided; Mean Difference (Final Values) = -.02, Standard Error of Mean .15
Statistical Analysis 3: Comparison: Screener Narrative vs Survivor Narrative; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Final Values) = .716, Standard Error of Mean .182

4. Secondary Outcome: Self-efficacy for Getting Screened for Colon Cancer
Description: Six items assess confidence in getting screened for colon cancer despite common barriers. Mean scores are created from response options that range from 1=not at all confident to 7=very confident. Higher scores reflect greater confidence in getting colorectal cancer screening. Means will be compared between all three study groups.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline survey, intervention, and immediate post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a 7-point response scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a 7-point response scale | 5.80 (1.36) | 5.81 (1.34) | 5.66 (1.33)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = 0.55, ANOVA; F-value = .608

5. Secondary Outcome: Affect
Description: Using the Positive and Negative Affect Schedule, we assessed the strength of 5 positive (happy, proud, strong, inspired, hopeful) and 5 negative (angry, guilty, sad, nervous, afraid) emotions felt during the assigned reading (1=Not at all - 7=Extremely). Higher mean subscale scores reflect stronger positive and negative emotions. Means will be compared between all three study groups.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline survey, intervention, and immediate post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a 7-point response scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a 7-point response scale
  Positive affect | 2.88 (1.58) | 3.22 (1.57) | 3.09 (1.47)
  Negative affect | 2.45 (1.34) | 2.07 (1.10) | 2.91 (1.41)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p < .001, ANOVA; F-value = 16.31
Statistical Analysis 2: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = 0.14, ANOVA; F-value = 2.00

6. Secondary Outcome: Defensive Information Processing
Description: Seven scales assessing defensive information processing will be assessed using previously validated measures for opt-out behavior (3 items), opt-out information (1 item), blunting (2 items), self-exemption (5 items), deny immediacy (3 items), counterarguing (4 items), and minimize the harm (2 items). Response options range from 1=strongly disagree to 7=strongly agree. Mean scores are created for each scale and higher scores reflect greater defensive information processing. Means will be compared between all three study groups.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline survey, intervention, and immediate post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a 7-point response scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a 7-point response scale
  Opt-out information | 2.79 (1.85) | 2.54 (1.68) | 2.90 (1.77)
  Opt-out behavior | 3.72 (1.75) | 3.69 (1.82) | 3.68 (1.85)
  Blunting | 3.75 (1.79) | 3.63 (1.68) | 3.78 (1.76)
  Self-exemption | 3.15 (1.75) | 3.30 (1.83) | 3.06 (1.77)
  Suppression | 2.97 (1.27) | 3.10 (1.33) | 2.83 (1.23)
  Counterarguing | 2.17 (1.13) | 2.31 (1.26) | 2.30 (1.36)
  Normalize the risk | 2.89 (1.39) | 2.87 (1.44) | 3.05 (1.55)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .19, ANOVA; F-value = 1.68
Statistical Analysis 2: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .98, ANOVA; F-value = .021
Statistical Analysis 3: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .73, ANOVA; F-value = .312
Statistical Analysis 4: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .496, ANOVA; F-value = .702
Statistical Analysis 5: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .154, ANOVA; F-value = 1.88
Statistical Analysis 6: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .514, ANOVA; F-value = .667
Statistical Analysis 7: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .514, ANOVA; F-value = .666

7. Secondary Outcome: Absolute Perceived Susceptibility to Colon Cancer
Description: Absolute perceived risk was assessed with three items: I am at risk for developing colorectal cancer, If I do not get screened regularly, I would feel vulnerable to developing colorectal cancer, If I do not get screened regularly, it is likely that I will develop colorectal cancer. Response options range from 1=strongly disagree to 5=strongly agree. Mean scale scores were created and higher scores reflect greater perceived susceptibility to colorectal cancer. Mean scores will be compared between all three study groups.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline survey, intervention, and immediate post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a 5-point response scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a 5-point response scale | 2.98 (0.76) | 3.03 (0.72) | 3.08 (0.78)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .56, ANOVA; F-value = .59

8. Other Pre Specified Outcome: Social Influence
Description: Social influence will be assessed with three items developed for this study based on standard measures that include physician, family, and friends as important social referents encouraging colorectal cancer screening. Response options range from 1=strongly disagree to 7=strongly agree. Mean scores were created and higher scores reflect greater perceived social influence for getting screened for colorectal cancer. Means will be compared between all three study groups.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline survey, intervention, and immediate post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a scale | 5.34 (1.33) | 5.40 (1.24) | 5.32 (1.19)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .84, ANOVA; F-value = .18

9. Other Pre Specified Outcome: Worry
Description: Worry was assessed with four items regarding worry about getting colorectal cancer, having a test that shows they have colorectal cancer, concern that colorectal cancer screening will be physically uncomfortable, and concern that there could be complications from the test. Response options ranged from 1=strongly disagree to 5=strongly agree. Mean scores were created (Range 1-5); higher scores reflect greater worry. Means will be compared between all three study groups.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline survey, intervention, and immediate post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a scale | 2.62 (0.99) | 2.66 (0.82) | 2.78 (1.01)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .31, ANOVA; F-value = 1.16

10. Other Pre Specified Outcome: Perceived Benefits and Barriers of Colorectal Cancer Screening
Description: Perceived colorectal cancer screening benefits (8 items) barriers (6 items) are assessed with items from previously validated scales. Response options range from 1=strongly disagree to 7=strongly agree. Mean scores were created for each scale; higher scores reflect greater perceived benefits and barriers of getting screened. Means will be compared between all three study groups.
Time Frame: Immediately post-intervention
Population: Participants who completed the baseline survey, intervention, and immediate post-intervention survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
Number analyzed (Participants) | 159 | 155 | 159
units on a scale
  Perceived benefits | 5.98 (0.92) | 6.08 (0.93) | 5.92 (1.00)
  Perceived barriers | 3.15 (1.34) | 3.15 (1.29) | 3.10 (1.34)
Statistical Analysis 1: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .31, ANOVA; F-value = 1.17
Statistical Analysis 2: Comparison: Information Only vs Screener Narrative vs Survivor Narrative; Test type: Superiority; p = .95, ANOVA; F-value = 0.056

ADVERSE EVENTS:
Time Frame: Participants were engaged in the study for approximately 12 months from baseline to final follow up survey.
Description: The only foreseeable adverse events that could arise from participation in the online study included negative affect including cancer worry as a result of reading about colorectal cancer risk, or a breach of confidentiality by researchers or hackers.
Arm/Group | Information Only | Screener Narrative | Survivor Narrative
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/155 | 0/159
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/155 | 0/159
Other Adverse Events (participants affected / at risk) | 0/159 | 0/155 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT02485561/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT02485561/ICF_001.pdf